CLINICAL TRIAL: NCT03625011
Title: Gabapentin Premedication to Reduce Postoperative Pain for Pediatric Tonsillectomy/Adenoidectomy: Randomized Control Trial
Brief Title: Gabapentin Premedication to Reduce Postoperative Pain for Pediatric Tonsillectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Margaret Gettis, Nurse Scientist, Children's Healthcare of Atlanta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IRB 18-052
Record Dates: First submitted 2018-07-20; First posted 2018-08-10 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Tonsillitis; Tonsillectomy
Keywords: Pain Relief; Non-Narcotic Pain relief
MeSH Terms: conditions — Tonsillitis | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants will be randomized to either Control Group or Gabapentin Group
  Interventions: Drug: Gabapentin
- Gabapentin Group (Active Comparator): Participants will be randomized to either Control Group or Gabapentin Group
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — This double blinded randomized control trial will enroll 50 children age 3-18 years, undergoing T/As. Patients will be receiving either one gabapentin dose (15mg/kg up to 600mg) or placebo preoperatively. Both control and test group will receive the standard narcotic regimen intraoperatively.
  Other Names: Neurontin

SUMMARY:
The purpose of this pilot study: 1) to examine the use of gabapentin in reducing pain in the first 48 hours postoperatively including the total amount of narcotics mg/kg given 2) to record the time to first analgesic postoperatively and 3) to compare Wong Baker and the 0-10 numeric pain distress scale scores at 12, 24 and 48 hours postoperatively. We hypothesize one 15mg/kg (up to 600mg) dose of gabapentin will decrease mean narcotic amounts in mg/kg compared to participants who do not receive preoperative gabapentin and will demonstrate a decreased mean time to first analgesic as well as to lower mean pain scores for each age group at 12, 24 and 48 hours.

DETAILED DESCRIPTION:
This double blinded randomized control trial will enroll 50 children age 3-18 years, undergoing T/As from a regional healthcare organization. Patients will be receiving either one gabapentin dose (15mg/kg up to 600mg) or placebo preoperatively. Both control and test group will receive the standard narcotic regimen intraoperatively. Additionally, young children will receive instruction for Tylenol and Motrin postoperatively while teenagers will receive a narcotic prescription. Outcome measurements include: mean Tylenol mg/kg, Motrin mg/kg and narcotic mg/kg use. Additional measurements: Mean time to first analgesic. Phone interviews with the research nurse for three days postoperatively will elicit pain scores at 12, 24 and 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* participants age 3-18 years
* ASA class 1 or 2
* elective Tonsillectomy/Adenoidectomy
* outpatient setting.

Exclusion Criteria:

* BMI >40kg/m2
* history of renal insufficiency, chronic pain
* allergy to gabapentin
* history of developmental delay

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Narcotic Consumption | First 48 hours postoperatively
  To examine the use of gabapentin in reducing pain in the first 48 hours postoperatively including the total amount of narcotics mg/kg(weight and height will be combined to report BMI in kg/m^2).

SECONDARY OUTCOMES:
First Analgesic Timing | First 48 Hours postoperatively
  To record the time to first analgesic postoperatively
Pain Scale Scores | 12, 24 and 48 hours postoperatively.
  To compare the Wong- Baker FACES Pain Rating Scale and the 1-10 numeric pain distress scale pain scores at 12, 24 and 48 hours postoperatively. The 0-10 Numeric Pain Distress Pain Scale utilizes number gradations to describe pain for school age children and adolescents. A zero score means the absence of pain while a five describes distressing pain and a ten infers unbearable pain. As for the Wong-Baker FACES Scale, a series of faces can be shown to children over the age of three. The six faces depict facial expressions with zero-no hurt at all, one-hurts just a little bit, two-hurts a little more, three-hurts even more, four-hurts a whole lot, and five- hurts as much as you can imagine. No subscales will be used or combined.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Calamaro, PhD, CPNP-PC, Study Chair — Institutional Review Board
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Amani S, Abedinzadeh MR. Effects of Oral Gabapentin, Local Bupivacaine and Intravenous Pethidine on Post Tonsillectomy Pain. Iran J Otorhinolaryngol. 2015 Sep;27(82):343-8. PMID 26568937
- [Background] Amin SM. Evaluation of gabapentin and dexamethasone alone or in combination for pain control after adenotonsillectomy in children. Saudi J Anaesth. 2014 Jul;8(3):317-22. doi: 10.4103/1658-354X.136417. PMID 25191179 (Retraction: PMID 30429763 Saudi J Anaesth. 2018 Oct-Dec;12(4):662)
- [Background] Amin SM, Amr YM. Comparison between preemptive gabapentin and paracetamol for pain control after adenotonsillectomy in children. Anesth Essays Res. 2011 Jul-Dec;5(2):167-70. doi: 10.4103/0259-1162.94758. PMID 25885382
- [Background] Hwang SH, Park IJ, Cho YJ, Jeong YM, Kang JM. The efficacy of gabapentin/pregabalin in improving pain after tonsillectomy: A meta-analysis. Laryngoscope. 2016 Feb;126(2):357-66. doi: 10.1002/lary.25636. Epub 2015 Sep 25. PMID 26404562
- [Background] Knipper E, Banta-Green CJ, Jimenez N. Opioid use disorder and misuse: A review of the epidemiology and medical implications for pediatric anesthesiologists. Paediatr Anaesth. 2017 Nov;27(11):1070-1076. doi: 10.1111/pan.13225. PMID 29030938
- [Background] Mohamed, M.H., Al-Sercy, H. (2014). Preoperative gabapentin decreases the incidence of postoperative vomiting and analgesic requirements after pediatric adenotonsillectomy. The Egyptian Journal of Otolaryngology. 225-228.
- [Background] Thiels CA, Anderson SS, Ubl DS, Hanson KT, Bergquist WJ, Gray RJ, Gazelka HM, Cima RR, Habermann EB. Wide Variation and Overprescription of Opioids After Elective Surgery. Ann Surg. 2017 Oct;266(4):564-573. doi: 10.1097/SLA.0000000000002365. PMID 28697049

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03625011/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03625011/ICF_001.pdf